CLINICAL TRIAL: NCT02879188
Title: Ambulation Versus Standing on Postoperative Day 0: A Randomized, Controlled Trial
Brief Title: Ambulation Versus Standing on Postoperative Day 0
Acronym: PT on POD 0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Craig J Della Valle, MD, Professor of Orthopaedic Surgery; Chief, Division of Adult Reconstructive Surgery, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1234568
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis
Keywords: degenerative joint disease; total knee arthroplasty; physical therapy; arthroplasty, replacement, knee
MeSH Terms: conditions — Osteoarthritis; Joint Diseases | interventions — Physical Therapy Modalities; Standing Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ambulation (Experimental): Patients will initiate inpatient physical therapy on the day of their surgery including attempted ambulation with an assistive device that is supervised by a physical therapist.
  Interventions: Other: Physical Therapy
- Standing (Active Comparator): Patients will initiate inpatient physical therapy on postoperative day 1. On the day of their surgery they will dangle their feet over the edge of the bed with supervision of nursing.
  Interventions: Other: Standing

INTERVENTIONS:
Other: Physical Therapy — Patients will initiate inpatient physical therapy on the day of their surgery including attempted ambulation with an assistive device that is supervised by a physical therapist.
  Arms: Ambulation
Other: Standing — Patients will initiate inpatient physical therapy on postoperative day 1. On the day of their surgery they will dangle their feet over the edge of the bed with supervision of nursing.
  Arms: Standing

SUMMARY:
The purpose of this study is to determine the impact of the timing of physical therapy (PT) initiation on postoperative length of stay and the time to physical therapy clearance following total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* scheduled for primary TKA (Total Knee Arthroplasty) for any degenerative condition
* Anesthesia for TKA is Spinal + Regional block (Adductor Canal Block)

Exclusion Criteria:

* require assistive devices (walker, wheelchair) for ambulation preoperatively
* planning to go to a subacute nursing facility or acute rehab facility following surgery
* < 18 yrs of age
* not willing to participate or unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2016-10; Primary Completion 2018-05 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Length of Hospitalization Stay | 5 days
  The length of time patients stay in the hospital will be recorded and compared between groups.

SECONDARY OUTCOMES:
Patient Satisfaction | 1 week
  Patients will be prospectively surveyed at discharge and asked questions about their satisfaction with their care during their hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Della Valle, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No